CLINICAL TRIAL: NCT05367999
Title: Development of a Clinical Decision Aid for the Differential Diagnosis of Transient Loss of Consciousness
Brief Title: A Clinical Decision Aid for Diagnosing Transient Loss of Consciousness
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH20060
Record Dates: First submitted 2022-04-19; First posted 2022-05-10 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Consciousness Disorder
Keywords: TLOC; Seizures; Epilepsy; Syncope
MeSH Terms: conditions — Consciousness Disorders; Seizures; Epilepsy; Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting with TLOC: A concurrent nested qualitative-quantitative design is used. Patients first presenting to an ED with TLOC (and witnesses) who have contributed to the quantitative part of this project will be offered participation in a qualitative interview study after completion of the iPEP during the initial study procedure. Capturing variation based on diagnosis, gender, age and participant/witness role, a purposive sample of participating participants and witnesses will be invited to semi-structured interviews in which they will be prompted to discuss their experiences of using the iPEP and their views on the accuracy in describing their peri-episodal experiences.
  Interventions: Diagnostic Test: initial Paroxysmal Event Profile

INTERVENTIONS:
Diagnostic Test: initial Paroxysmal Event Profile — The initial Paroxysmal Event Profile (iPEP) was derived from the paroxysmal event profile (PEP) and paroxysmal event observer (PEO) to provide a diagnostic tool aiming to differentiate between the most common underlying reasons for TLOC presentations: syncope, epilepsy, and dissociative seizures. The iPEP is a 35-item questionnaire developed from the PEP and PEO.5,25 The 5-point frequency scales used in response to each symptom in the PEP and PEO have been replaced with a binary 'present'/'not present' classification in recognition of the fact that the target patient group may have experienced only one or a few episodes of TLOC.

SUMMARY:
BACKGROUND: Transient loss of consciousness (TLOC) - defined as spontaneous disruption of consciousness not due to head trauma and with complete recovery - has a lifetime prevalence of 50%. It is one of the commonest neurological complaints in primary and emergency care. Over 90% of TLOC is due to either syncope, epilepsy or dissociative seizures (DS, also known as 'Psychogenic Nonepileptic Seizures'). The rapid and accurate distinction of these diagnoses is vital to allow appropriate further management but at least 20-30% of patients are not managed optimally or misdiagnosed. We have previously demonstrated that, in patients with established diagnoses of epilepsy, syncope, or DS, an automated classifier using only information from 36 questions based on patient experience and lay witness reports (the initial Paroxysmal Event Profile, iPEP) could accurately diagnose 86.0% of patients (with 100% sensitivity and 91.7% specificity for syncope)

AIMS: To calibrate the iPEP for discrimination between syncope, epilepsy, and DS in patients newly presenting with TLOC, validate its performance in an independent sample, and to explore acceptability of the use of such a tool to people with TLOC and witnesses.

METHODS: Nested qualitative-quantitative prospective single-centre development and validation of the iPEP in patients presenting to Emergency Departments, syncope or epilepsy clinics with first presentations of TLOC, with semi-structured interviews conducted with a purposive sample of participants from the quantitative study. The iPEP will be calibrated using a previously-described procedure for variable selection and training of Random Forest (RF) classifiers, and validated with assessment of overall classification accuracy, alongside sensitivity, specificity, positive and negative predictive values, and area under receiver-operating curve for each of the three target diagnoses. Performance will be evaluated against a benchmark set by results from previous research in patients with established diagnoses of epilepsy, syncope, and DS.

OUTPUTS: Results will be submitted for publication in academic and professional literature. If performance from feasibility can be replicated in validation, the iPEP will be suitable to begin process of registration as a medical device for implementation in clinical pathways to minimise inappropriate referrals and treatment, streamline patient pathways, and enable earlier ordering of appropriate investigations to ensure prompt and appropriate diagnosis and management. If pilot performance could be replicated in this population and proportional savings from current estimated costs of misdiagnosis achieved, this could potentially save £63.9 million of annual UK healthcare expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Patients first presenting with TLOC
* Referred to secondary care for diagnostic evaluation OR given firm diagnosis of syncope in accordance with European Society of Cardiology guidelines for syncope presentations not requiring further investigation
* Adult over the age of 16 years
* Able to complete iPEP questionnaire independently
* Participants do not need to be native English speaker but do need to have sufficient English language ability to complete iPEP without support

Initial Exclusion Criteria:

* Unable to give informed consent to participation in research
* Unable to complete iPEP independently
* Previous specialist (neurological or cardiological) assessment of TLOC

Criteria for exclusion from analysis:

* No firm clinical diagnosis of TLOC (and its cause) at end of 6-month follow-up period
* Mixed diagnosis of multiple TLOC-causing disorders at end of 6-month follow-up; we exclude these participants from analysis as they would not have a single reference standard diagnosis, thus their inclusion in development may reduce model performance (since their questionnaire answers will describe multiple different kinds of episode), and in validation there is no principled way to assess performance of the prediction model if they have more than one reference diagnosis. A previous study of patients with suspected seizures in this population found that only 1.1% of patients could not be given a single aetiological diagnosis, so we do not anticipate this resulting in many exclusions.4
* Evidence of previous specialist (neurological or cardiological) assessment of TLOC.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of screened admissions to the Emergency Department and Acute Medical Unit presenting with TLOC, as well as all new patients referred to the Neurology and Cardiology departments with TLOC.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
AUC for syncope | 6 months post-presentation
  We will compare classifier-predicted diagnoses against final diagnoses obtained by expert consensus review of medical records. We will define performance in terms of AUC for cardiogenic syncope.

SECONDARY OUTCOMES:
Overall classifier accuracy | 6 months post-presentation
  We will compare classifier-predicted diagnoses against final diagnoses obtained by expert consensus review of medical records. We will define performance in terms of classifier accuracy, and sensitivity, specificity, positive and negative predictive values for other diagnoses (i.e., epileptic/dissociative seizures). This will enable direct comparison with current rates of misdiagnosis.

OTHER OUTCOMES:
Participant experience | 6-month follow-up
  A purposive sample of participants who have consented to be contacted about the additional interview study will be invited to participate in the nested qualitative research. Those consenting will take part in a semi-structured interview by telephone or in person. To help inform future adaptation and implementation of the iPEP, participants' feedback and views on how to communicate the decision aid results will be explored. All interviews will be audio-recorded and transcribed verbatim. The data will be analysed using NVivo, and thematic analysis undertaken to identify recurring views and opinions.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Reuber, Principal Investigator — Honorary Consultant Neurologist; Alistair Wardrope, Principal Investigator — Specialty Registrar in Neurology
Locations (2):
- United Kingdom (2):
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Northern General Hospital, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: No